CLINICAL TRIAL: NCT03061552
Title: Influence of Dry Weight Adjustment by Inferior Vena Cava Sonography in Hemodialysis Patients on Quality of Life During Treatment
Brief Title: Inferior Vena Cava Sonography in Hemodialysis Patients and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 032416-HMO-CTIL
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2020-12

CONDITIONS: Hemodialysis Complication; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVCD arm (Experimental): IVCD-assisted determination of target post-dialysis weight
  Interventions: Diagnostic Test: sonographic measurement of inferior vena cava diameter
- conventional arm (No Intervention): conventional determination of target post-dialysis weight

INTERVENTIONS:
Diagnostic Test: sonographic measurement of inferior vena cava diameter — pre-dialysis measurement of inferior vena cava diameter using echocardiography
  Arms: IVCD arm

SUMMARY:
Determination of dry weight in patients with end-stage renal disease treated with hemodialysis is an unmet challenge in clinical nephrology. Current methods are imprecise, and thus many patients are hype- or hypovolemic, and suffer respective consequences such as hypertension, pulmonary congestion, cardiac hypertrophy, chronic dehydration, hypotension and shock.

Several techniques have been proposed to asses hydration status in dialysis patient, among them measurement of bioimpedance and biochemical markers. Sonographic measurement of the inferior vena cava diameter (IVCD) is a method under investigation for assessing hydration status. It is available, inexpensive and efficient, yet operator-dependent. In a single-center, blinded and controlled trial it has been shown to improve clinical outcomes in patients receiving hemodialysis.

In this study, we aim to assess the applicability and clinical utility of this method in our dialysis units. A crossover design is intended to examine the effect of IVCD measurement on quality of life and rate of hemodynamic adversities as compared with traditional estimation of dry weight.

DETAILED DESCRIPTION:
Introduction Patients with end-stage renal disease (ESRD) cannot regulate their fluid balance, and are dependent on dialysis for fluid removal. Fluid removal is dependent upon estimation of dry weight. Dry weight is defined as the post-dialysis weight under which a patient suffers (more often than not) from symptoms of hypotension. Today, clinical estimation of dry weight is based on physical examination. This method is inaccurate, and many patients suffer from the consequences of over- or under-estimation of their dry weight. Overestimation leads to hypertension, edema and pulmonary congestion, cardiac hypertrophy and failure. Underestimation results in chronic dehydration, hypotension, dizziness, muscle spasms, gastrointestinal disturbances, tinnitus and shock. Both over- and underestimation diminish quality of life. One of the methods proposed as objective estimators of hydration status is sonographic measurement of the inferior vena cava diameter (IVCD). Cheriex et al have determined that IVCD correlates with right atrial filling, and suggested that IVCD above 11.5 mm/m2 indicates hypervolemia, and values less than 8 mm/m2 indicate hypovolemia. Chang et al reported the only randomized controlled trial to examine quality of life and clinical outcomes of hemodialysis patients in whom IVCD was measured compared to patients in whom dry weight estimation was based solely on physical examination. They found lesser clinical mishaps and improved quality of life in the intervention group, an effect which was more pronounced in patients found to be hypovolemic. As this is the only reported randomized intervention, conducted with Asian participants, we sought to conduct a similar study in an independent hemodialysis population.

Objective Examination of the quality of life consequences of dry weight estimation in ESRD patients receiving dialysis with sonographic IVCD measurement.

Hypothesis We assume that adjustment of dry weight in ESRD patients receiving hemodialysis using sonographic IVCD measurements will improve quality of life.

Methods Study design: single-blinded cross-over clinical trial Study population: ESRD patients receiving chronic dialysis at the Hadassah Medical Center hemodialysis units. Exclusion criteria: pregnant women; patients treated with hemodialysis less than 3 months; significant tricuspid regurgitation; severe heart failure; patients with inadequate sonographic window for IVCD visualization.

Quantitative outcomes: Primary - rate of symptomatic hypotensive events during hemodialysis sessions; secondary - (1) quality of life, as evaluated using Short Form (SF)-36 questionnaire; (2) intradialysis clinical events: hypotensive episodes, gastrointestinal complaints, muscle spasm, tinnitus, headache and chest pain; (3) rate of emergent (unplanned) hemodialysis treatments; (4) average 24 h ambulatory blood pressure and sleep-related dipping.

Experimental methods: hemodialysis patients undergo monthly clinical evaluation by their primary nephrologist, including history, review of peri-dialysis blood pressure, physical examination and routine labs - which are basis for the monthly adjustment of target dry weight. Measurement of IVCD index will be performed twice in each participant, at the beginning of months 1 and 3, prior to the monthly visit by the primary nephrologist. Measurement will be performed as described by Cheriex et al. The primary nephrologist will be notified of the IVCD index performed at the beginning of month 3, and will be requested to adjust target post-dialysis weight accordingly. Participants will be blinded as to whether to not the primary nephrologist has been notified of the measurement.

Assessment of quality of life: self report by patients using SF-36 medical outcome study short form health survey scoring system, at the end of months 2 and 4.

Ambulatory blood pressure monitoring: will be performed using Oscar-2 devices (SunTech) at the ends of months 2 and 4.

Sample size analysis: calculation of sample size was guided by the primary outcome. We estimated that 4 hypotensive episodes occur across 14 monthly dialysis sessions, and that an intervention can reduce the number of episodes to 2 per 14 session. With a difference of 2 episodes and standard deviation of 2 episodes, alpha level of 0.05 and 90% power, with a 2-sided paired t-test sample size is 13 paired assessments (13 patients) (WINPEPI). Assuming incomplete followup, we intend to recruit up to 20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult ESRD patients receiving hemodialysis at the Hadassah Medical Center

Exclusion Criteria:

* Pregnant women; patients treated with hemodialysis less than 3 months; significant tricuspid regurgitation; severe heart failure; inadequate sonographic window for IVCD visualization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
symptomatic hypotension | 2 months
  rate of symptomatic hypotensive episodes during hemodialysis sessions per participant per month

SECONDARY OUTCOMES:
self-reported quality of life | 2 months
  self-reported quality of life using SF-36 questionnaire
intra-dialysis clinical events | 2 months
  rate of events: asymptomatic hypotension; gastrointestinal upset; muscle spasm; tinnitus; headache; chest pain
unplanned hemodialysis | 2 months
  rate of emergency hemodialysis treatments
interdialysis ambulatory blood pressure | 2 months
  interdialysis 24 h ambulatory blood pressure (ABPM)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah - Hebrew University Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang ST, Chen CL, Chen CC, Hung KC. Clinical events occurrence and the changes of quality of life in chronic haemodialysis patients with dry weight determined by echocardiographic method. Int J Clin Pract. 2004 Dec;58(12):1101-7. doi: 10.1111/j.1742-1241.2004.00124.x. PMID 15646404
- [Background] Cheriex EC, Leunissen KM, Janssen JH, Mooy JM, van Hooff JP. Echography of the inferior vena cava is a simple and reliable tool for estimation of 'dry weight' in haemodialysis patients. Nephrol Dial Transplant. 1989;4(6):563-8. PMID 2507979
- [Background] Abramson JH. WINPEPI updated: computer programs for epidemiologists, and their teaching potential. Epidemiol Perspect Innov. 2011 Feb 2;8(1):1. doi: 10.1186/1742-5573-8-1. PMID 21288353